CLINICAL TRIAL: NCT06396858
Title: A 2 x 2 Factorial Randomized Clinical Trial Evaluating Anti-inflammatory and Anti-thrombotic Strategy in Acute Ischemic Stroke
Brief Title: Anti-inflammatory and Anti-thrombotic Therapy With colcHicine and Low Dose Rivaroxaban for Major Adverse Cardiovascular Events Reduction in Ischemic Stroke
Acronym: ARCHIMEDES
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Brazilian Clinical Research Institute (Other)
Collaborators: Alliança Diagnostic (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 001/2023
Record Dates: First submitted 2024-01-04; First posted 2024-05-02 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Ischemic Stroke
Keywords: Stroke; Anticoagulation; rivaroxaban; colchicine
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Rivaroxaban; Colchicine

STUDY DESIGN:
Intervention Model Description: they will be randomized, simultaneously, in a 1:1 ratio, to rivaroxaban 2.5 mg BID or placebo, and colchicine 0.5 mg QD versus placebo, in a 2x2 factorial design. Therefore, the study will have four possible groups: rivaroxaban 2.5 mg BID + colchicine 0.5 mg QD; rivaroxaban 2.5 mg BID + colchicine placebo QD; rivaroxaban placebo BID + colchicine 0.5 mg QD; or rivaroxaban placebo BID + colchicine placebo QD
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Matching placebos will be produced for rivaroxaban and colchicine.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Active Comparator): rivaroxaban 2.5 mg Twice a day (BID) + colchicine 0.5 mg once daily (QD)
  Interventions: Drug: Rivaroxaban 2.5 Mg Oral Tablet; Drug: Colchicine 0.5 MG
- Group 2 (Active Comparator): rivaroxaban 2.5 mg BID + colchicine placebo QD
  Interventions: Drug: Rivaroxaban 2.5 Mg Oral Tablet; Drug: Placebo Colchicine
- Group 3 (Active Comparator): rivaroxaban placebo BID + colchicine 0.5 mg QD
  Interventions: Drug: Colchicine 0.5 MG; Drug: Placebo Rivaroxaban
- Group 4 (Placebo Comparator): rivaroxaban placebo BID + colchicine placebo QD
  Interventions: Drug: Placebo Rivaroxaban; Drug: Placebo Colchicine

INTERVENTIONS:
Drug: Rivaroxaban 2.5 Mg Oral Tablet — Patients will receive one tablet, per oral or orogastric route, twice a day, for a maximum of 12 months.
  Other Names: Xarelto
  Arms: Group 1; Group 2
Drug: Colchicine 0.5 MG — Patients will receive one tablet, per oral or orogastric route, once a day, for a maximum of 12 months.
  Other Names: Colchis
  Arms: Group 1; Group 3
Drug: Placebo Rivaroxaban — Patients will receive one tablet, per oral or orogastric route, twice a day, for a maximum of 12 months.
  Arms: Group 3; Group 4
Drug: Placebo Colchicine — Patients will receive one tablet, per oral or orogastric route, once a day, for a maximum of 12 months.
  Arms: Group 2; Group 4

SUMMARY:
The ARCHIMEDES study (Anti-inflammatory and anti-thRombotic therapy with colCHicine and low dose rIvaroxaban for Major adverse cardiovascular Events reDuction in ischEmic Stroke) will be a randomized, double-blind, 2x2 factorial clinical trial, which will include at least 3000 and up to a maximum of 4500 patients with ischemic stroke without indication of oral anticoagulation.

DETAILED DESCRIPTION:
In patients with ischemic stroke, within 14 days of symptom onset, to establish the efficacy and safety of two strategies in parallel: low-dose rivaroxaban and low-dose colchicine, compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute ischemic stroke aged ≥18 years old who, regardless of etiology and mechanism, do not have a definitive indication for anticoagulation, and whose symptoms onset has been within the last 14 days;
* Receiving standard therapy for acute management of ischemic stroke;
* For patients treated with fibrinolytics, a minimum period of 24 hours after the infusion of the lytic drug is required for randomization into the study.

Exclusion Criteria:

* Modified Rankin score of 4 or more at randomization;
* Refusal to provide consent;
* Severe renal failure, with glomerular filtration rate (by CKD-EPI) estimated at <15 mL/min/1.73 m2;
* Severe liver failure (child C);
* Indication for full-dose anticoagulation (for example, venous thromboembolism or atrial fibrillation);
* Previous hemorrhagic stroke or history of intracranial hemorrhage;
* Systemic treatment with a potent CYP 3A4 inhibitor (such as azole antifungals and protease inhibitors), or with a potent 3A4 inducer (such as rifampicin, phenytoin, phenobarbital, or carbamazepine);
* History of inflammatory bowel disease or chronic diarrhea;
* Prolonged treatment (> 1 month) with immunosuppressants or systemic corticosteroids;
* History of recurrent pneumonia (3 or more hospitalizations in the last 12 months);
* Pregnancy or breastfeeding;
* Any other comorbidity other than stroke and CV disease (e.g., metastatic cancer) that, in the investigator's opinion, has a significant impact on the 12-month survival.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4500 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy endpoint: Time to cardiovascular death, stroke, myocardial infarction (MI), or urgent arterial | 12 months
  Time to cardiovascular death, stroke, myocardial infarction (MI), or urgent arterial revascularization
Primary safety endpoint (rivaroxaban versus placebo): Time to major bleeding according to the International Society of Thrombosis and Hemostasis classification | 12 months
  Time to major bleeding according to the International Society of Thrombosis and Hemostasis classification
Primary safety endpoint (colchicine versus placebo): Hospitalization for respiratory infections | 12 months
  Time to first hospitalization for respiratory infections

SECONDARY OUTCOMES:
Time to fatal or non-fatal stroke | 12 months
  Time to fatal or non-fatal stroke
Time to CV death, MI, or stroke | 12 months
  Time to CV death, MI, or stroke
Time to death from all causes, MI, or stroke | 12 months
  Time to death from all causes, MI, or stroke
Time to fatal or non-fatal stroke, death, or transient ischemic attack | 12 months
  Time to fatal or non-fatal stroke, death, or transient ischemic attack
Net clinical endpoint: time to CV death, MI, stroke, fatal bleeding, or critical site bleeding | 12 months
  Time to CV death, MI, stroke, fatal bleeding, or critical site bleeding
Time to all-cause death | 12 months
  Time to all-cause death

OTHER OUTCOMES:
modified Rankin score | 12 months
  modified Rankin score as ordinal outcome
Venous thromboembolism | 12 months
  Time to first venous thromboembolism
New-onset atrial fibrillation | 12 months
  time to new-onset atrial fibrillation
Microvascular obstruction at head MRI (substudy) | 12 months
  Microvascular obstruction at head MRI (substudy)

CONTACTS AND LOCATIONS:
Overall Officials: Renato D Lopes, MD, PhD, Study Chair — Brazilian Clinical Research Institute